CLINICAL TRIAL: NCT04650321
Title: Evaluating the Feasibility of Pandemic Forward, Telehealth Based Home Based Infusions
Brief Title: Home Based Infusions for Ocrelizumab
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-2153
Record Dates: First submitted 2020-11-16; First posted 2020-12-02 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Single arm clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Home infusion of ocrelizumab (Experimental): Patients will receive infusion of ocrelizumab at home, instead of at clinic.
  Interventions: Drug: Ocrelizumab at home

INTERVENTIONS:
Drug: Ocrelizumab at home — Patients will receive ocrelizumab infusion at home.

SUMMARY:
The goal is to assess the safety and effectiveness of home ocrelizumab infusion.

DETAILED DESCRIPTION:
The safety of home ocrelizumab infusion will be assessed by monitoring for infusion reactions and adverse events, and comparing proportions/rates to existing studies. Patient reported outcomes (PROs) will compare pre to post infusion.

ELIGIBILITY:
Inclusion Criteria:

* Current active patient of Rocky Mountain MS Center at the time of final study consent.
* Between 18-55 years of age at the time of final study consent.
* Diagnosis of primary progressive or relapsing MS as defined by the 2017 McDonald criteria.19
* Has at minimum completed their first 600 mg dose of ocrelizumab.
* Is physically residing in the Denver metro, Fort Collins or Colorado Springs area at the time of final study consent.
* Has a Patient Determined Disease Steps (PDDS) between 0 to 6.5 20
* Can complete patient reported outcomes developed and validated as English written scales.
* Must be able and willing to give meaningful, informed consent via electronic signature prior to participation in the study, in accordance with local and FDA regulatory requirements.
* Whose treating neurologist at the RMMSC feels that continuing ocrelizumab s medically appropriate based on at the time of final study consent.

Exclusion Criteria:

* Not pregnant, intentions to get pregnant or lactating at the time of final study consent and on the day of infusion.
* Has previously not participated in the SaROD trial at the RMMSC site.
* Any of the following abnormal laboratory results as processed by a University of Colorado Hospital laboratory site and deemed clinically inappropriate to proceed with a home infusion by the treating neurologist at RMMSC.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Severe infusion reactions | 24 hours after infusion
  Proportion of patients with infusion reactions greater than or equal to 3 on the National Cancer Institute's Common Terminology
Infusion reactions | 24 hours after infusion
  Proportion of patients with infusion reactions greater than or equal to 1 on the National Cancer Institute's Common Terminology

SECONDARY OUTCOMES:
Severe infusion reactions compared to historic controls. | 24 hours after infusion
  Difference in proportion of patients with infusion reactions greater than or equal to 3 on the National Cancer Institute's Common Terminology between home infusion and the CHORDS and ENSEMBLE historical controls.
Infusion reactions compared to historic controls. | 24 hours after infusion
  Difference in proportion of patients with infusion reactions greater than or equal to 1 on the National Cancer Institute's Common Terminology between home infusion and the CHORDS and ENSEMBLE historical controls.
Validated Patient Reported Outcomes (PROs) - PROMIS 10 Physical | 2 months
  Change in PROMIS 10 values between pre and post infusion. Ranges from 10 to 50. Higher numbers indicate better well being.
Validated Patient Reported Outcomes (PROs) - PROMIS 10 Mental | 2 months
  Change in PROMIS 10 values between pre and post infusion. Ranges from 10 to 50. Higher numbers indicate better well being.
Validated Patient Reported Outcomes (PROs) - Neuro-QOL Anxiety | 2 months
  Change in Neuro-QOL Anxiety values between pre and post infusion. Score is transformed to a T score, with population mean of 50 and population standard deviation of 10. T score can range from 36.4 to 76.8. Higher scores mean more anxiety, and hence worse.
Validated Patient Reported Outcomes (PROs) - Neuro-QOL Depression | 2 months
  Change in Neuro-QOL Depression values between pre and post infusion. Score is transformed to a T score, with population mean of 50 and population standard deviation of 10. T score can range from 36.9 to 75.0. Higher scores mean more depression, and hence worse.
Validated Patient Reported Outcomes (PROs) - Patient Determined Disease Steps (PDDS) | 2 months
  Change in PDDS values between pre and post infusion.
Adverse events | 2 months
  Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Timothy L Vollmer, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Amerita, Centennial, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vollmer TL, Cohen JA, Alvarez E, Nair KV, Boster A, Katz J, Pardo G, Pei J, Raut P, Merchant S, MacLean E, Pradhan A, Moss B. Safety results of administering ocrelizumab per a shorter infusion protocol in patients with primary progressive and relapsing multiple sclerosis. Mult Scler Relat Disord. 2020 Nov;46:102454. doi: 10.1016/j.msard.2020.102454. Epub 2020 Aug 18. PMID 33045496